CLINICAL TRIAL: NCT04864340
Title: Crossover Randomized Clinical Trial to Evaluate the Effectiveness and Safety of Pupillometry as an Objective Measurement of Nociception in Healthy Volunteers.
Brief Title: Clinical Trial Using Pupillometry to Measure Nociception in Healthy Volunteers.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: IIBSP-PUP-2019-01
Record Dates: First submitted 2021-04-13; First posted 2021-04-28 (Actual); Last update posted 2021-05-19 (Actual); Status verified 2021-05

CONDITIONS: Nociceptive Pain; Pupillary Light Reflex Lost; Healthy; Pain, Procedural; Gender; Anxiety
MeSH Terms: conditions — Nociceptive Pain; Pain, Procedural; Coitus; Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- threshold stimulation (tetanic) (Experimental)
  Interventions: Device: CE marked medical device
- upper threshold stimulation (tetanic) (Experimental)
  Interventions: Device: CE marked medical device
- threshold stimulation (pressure) (Experimental)
  Interventions: Device: Algometer
- upper threshold stimulation (pressure) (Experimental)
  Interventions: Device: Algometer
- non nociceptive procedure (fine touch) (Placebo Comparator)
  Interventions: Procedure: Comparator

INTERVENTIONS:
Device: CE marked medical device — Tetanic stimulation
  Arms: threshold stimulation (tetanic); upper threshold stimulation (tetanic)
Device: Algometer — Pressure stimulation
  Arms: threshold stimulation (pressure); upper threshold stimulation (pressure)
Procedure: Comparator — Non-nociceptive procedure (fine touch)
  Arms: non nociceptive procedure (fine touch)

SUMMARY:
Pupillometry has been used in healthy volunteers to investigate the usefulness of the pupil light reflex as an indicator of pain intensity on pressure as a nociceptive stimulus. In this sense, it is necessary to check if the pupillometry is sensitive to different types or sources of pain. One of these devices is the Algiscan® portable pupillometer (IdMed, Marseille, France), which we propose to use in the present study. This pupillometer has previously been used in healthy volunteers, and in patients admitted to the intensive care unit, subjected to mechanical ventilation and sedation / analgesia.

This study in healthy volunteers aims to evaluate whether the PDR can be a reliable and discriminatory measure of the intensity of nociception, applying various types of nociceptive stimuli. If so, this study could lead to the use of pupillometry as an objective measure of nociception in settings where patients cannot communicate, such as intensive care areas or perioperative settings.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects of both sexes (balanced)
2. Caucasian race
3. Ages between 25 and 65 years old (balanced, 50% from 25-45 and 50% from 45-65)
4. Body weight within the normal range (Quetelet index: 19-30)
5. Clinical history, physical examination and vital signs within normality
6. Free acceptance to participate, with written informed consent

Exclusion Criteria:

1. Previous history of alcoholism or drug dependence (year prior to the screening visit or daily alcohol consumption> 40 gr / day for men or> 24 gr / day for women)
2. Significant consumption of stimulating drinks (> 5 coffees, teas, chocolate or cola drinks / day).
3. Taking any medication in the 15 days prior to the study and / or medicinal plants that may have an effect on the pupil (beta-blockers, droperidol, metoclopramide, clonidine ...). Oral contraceptives and paracetamol will be allowed.
4. Pregnancy (β-hCG test).
5. Menstruation and / or dysmenorrhea on the day of the study
6. Family or personal history or clinical evidence of psychiatric, neurological or ophthalmological problems: anxiety, depression, Parkinson's, glaucoma, dry eyes, retinal diseases, eye surgery and pupil abnormalities, presenting migraine pathology and diabetes
7. Pupillary diameter ≥ 5mm
8. Smokers or ex-smokers <6 months.
9. Have participated in a clinical trial in the 3 months prior to the start of this study.

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 30 (Estimated)
Dates: Start 2021-04-30 (Actual); Primary Completion 2021-05 (Estimated); Study Completion 2021-05 (Estimated)

PRIMARY OUTCOMES:
Change in Pupillary Dilatation Reflex (PDR) | Change in Pupillary Dilatation Reflex (PDR) from baseline to +10 minutes (with non-nociceptive procedure (fine touch))
  Measure of Pupillary Dilatation Reflex (PDR) in % obtained by AlgiScan®
Change in Pupillary Dilatation Reflex (PDR) | Change in Pupillary Dilatation Reflex (PDR) from baseline to 20 minutes after tetanic stimulation (by Algiscan®)
  Measure of Pupillary Dilatation Reflex (PDR) in % obtained by AlgiScan® after tetanic stimulation (by Algiscan®)
Change in Pupillary Dilatation Reflex (PDR) | Change in Pupillary Dilatation Reflex (PDR) from baseline to 30 minutes after tetanic stimulation (by Algiscan®)
  Measure of Pupillary Dilatation Reflex (PDR) in % obtained by AlgiScan® after tetanic stimulation (by Algiscan®)
Change in Pupillary Dilatation Reflex (PDR) | Change in Pupillary Dilatation Reflex (PDR) from baseline to 40 minutes after tetanic stimulation (by Algiscan®)
  Measure of Pupillary Dilatation Reflex (PDR) in % obtained by AlgiScan® after tetanic stimulation (by Algiscan®)
Change in Pupillary Dilatation Reflex (PDR) | Change in Pupillary Dilatation Reflex (PDR) from baseline to 50 minutes after tetanic stimulation (by Algiscan®)
  Measure of Pupillary Dilatation Reflex (PDR) in % obtained by AlgiScan® after tetanic stimulation (by Algiscan®)

SECONDARY OUTCOMES:
Change in Pupillary Dilatation Reflex (PDR) | Change in Pupillary Dilatation Reflex (PDR) from baseline to + 60 minutes after pressure estimulation
  Measure of Pupillary Dilatation Reflex (PDR) in % obtained by AlgiScan® after pressure estimulation (by algometer Somedic®)
Change in Pupillary Dilatation Reflex (PDR) | Change in Pupillary Dilatation Reflex (PDR) from baseline to +70 minutes after pressure estimulation
  Measure of Pupillary Dilatation Reflex (PDR) in % obtained by AlgiScan® after pressure estimulation (by algometer Somedic®)
Change in Pupillary Dilatation Reflex (PDR) | Change in Pupillary Dilatation Reflex (PDR) from baseline to +80 minutes after pressure estimulation
  Measure of Pupillary Dilatation Reflex (PDR) in % obtained by AlgiScan® after pressure estimulation (by algometer Somedic®)
Change in Pupillary Dilatation Reflex (PDR) | Change in Pupillary Dilatation Reflex (PDR) from baseline to +90 minutes after pressure estimulation
  Measure of Pupillary Dilatation Reflex (PDR) in % obtained by AlgiScan® after pressure estimulation (by algometer Somedic®)

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital de la Santa Creu i Sant Pau, Barcelona, Spain